CLINICAL TRIAL: NCT07326228
Title: Effect of Combined Inspiratory Muscle Training and Aerobic Exercises on Ventilatory Function in Adults With Repaired Tetralogy of Fallot
Brief Title: Effect of Exercises on Ventilatory Function in Adult With TOF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Ahmed Khalaf Ismail, Physical Therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/005997
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Tetralogy of Fallot (TOF); Adults With Repaired Tetralogy of Fallot
Keywords: congenital heart disease; tetralogy of Fallot; inspiratory muscle training; aerobic exercise; ventilatory functions; functional capacity; Quality of life
MeSH Terms: conditions — Tetralogy of Fallot; Heart Defects, Congenital | interventions — Exercise; Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined respiratory muscle training and aerobic training (Experimental): participants will receive respiratory muscle training via threshold IMT device in addition to moderate intensity aerobic exercise
  Interventions: Other: aerobic exercise; Other: respiratory muscle training
- aerobic exercise (Active Comparator): participants will receive moderate intensity aerobic exercise
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise — moderate intensity aerobic exercises on a treadmill:
  * Symptom-limited treadmill exercise training will be carried out at baseline for each participant following the modified Bruce protocol to estimate each participant's peak heart rate.
  * the target heart rate during training will be 50-60 % of each participant's heart rate reserve (moderate intensity exercise)
  * each session will have 5-10 min warm up, at least 20 min of moderate intensity aerobic exercise , and 5-10 min of cool down
Other: respiratory muscle training — respiratory muscle training via threshold inspiratory muscle trainer (IMT) device:
  * maximum inspiratory effort will be detected for each participant as the maximum resistance at which the participant can efficiently achieve 10 breathing cycles, via (Threshold IMT device)
  * the training will be initiated with a low-intensity load (20-30%) of the participant's maximum inspiratory effort via (Threshold IMT device). Then, the intensity will increase gradually by 5% according to the participant's tolerance weekly until achieving 50% of maximum inspiratory effort.
  * the session will be formed of six sets, each set consisting of five deep breaths against the (Threshold IMT device), with a short interval of 1-2-minute rest between sets.
  Other Names: Threshold inspiratory muscle training; inspiratory muscle training
  Arms: combined respiratory muscle training and aerobic training

SUMMARY:
The goal of this clinical trial is to learn if combined inspiratory muscle training and aerobic exercise can improve ventilatory function in adults with repaired Tetralogy of Fallot (TOF). It will also learn if exercises work to raise functional capacity and Quality of life (QoL) . The main questions it aims to answer is:

* Dose combined inspiratory muscle training and aerobic exercise (study group) improve ventilatory function in adults with repaired (TOF) more than aerobic exercise only (control group)?
* Can combine inspiratory muscle training and aerobic exercise (study group) raise functional capacity and (QoL) in adults with repaired (TOF) more than aerobic exercise only (control group)?

Researchers will compare between combination of inspiratory muscle training and aerobic exercise on one group and the aerobic exercise only on other group, on ventilatory function, functional capacity and (QoL) on adults with repaired TOF.

Participants will:

On study group , participants will perform respiratory muscle training in addition to moderate intensity aerobic exercise for 6 weeks. 3 times/week

On controlled group , participants will perform moderate intensity aerobic exercise for 6 weeks. 3 times/week.

all participants will test ventilatory function , functional capacity and will answer a survey questions about their quality of life before and after training

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with TOF.
* Have surgical correction of the abnormality.
* Class II-III according to New York Heart Association (NYHA)
* Ejection fracture > 40
* Vitally stable during the study period

Exclusion Criteria:

* Resent cardiopulmonary surgery or intervention "less than 6 months"
* Presence of pulmonary disease which is not a complication of TOF (eg:

bronchial asthma, lung fibrosis…..)

* Neuromuscular or musculoskeletal disease and severe scoliosis affecting pulmonary function or physical exercise.
* Mental or physical limitations
* active infection or systemic illness.
* Hemodynamic instability
* Mouth burn, injury, or deformities
* Implanted pacemaker

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
"Change from Baseline in Ventilatory function : Forced vital capacity (FVC) , Forced expiratory volume in 1 second (FEV1), expiratory vital capacity (EVC) and inspiratory vital capacity (IVC). | At Baseline and after 6 weeks of training

SECONDARY OUTCOMES:
Change from Baseline in Six-minute walk test (6MWT) | At Baseline and after 6 weeks of training
changes from baseline in 36-Item Short Form Health Survey (SF-36) | at Baseline and after 6 weeks of training
  as an assessment of quality of live

IPD SHARING:
Plan to Share IPD: Undecided